CLINICAL TRIAL: NCT04724577
Title: Phase I Study on Carbon Ion Radiotherapy in 12 Fractions for Localized Prostate Cancer
Brief Title: 12 Fractions Carbon Ion Radiotherapy for Localized Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Ping Li, Principal Investigator, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PCa2019-01
Record Dates: First submitted 2021-01-23; First posted 2021-01-26 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Radiotherapy; Prostate Cancer
Keywords: localized prostate cancer; carbon ion radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Intervention Model Description: dose escalation study for carbon ion radiotherapy in prostate cancer
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carbon ion treatment (Experimental): dose escalation study with five dose levels [54GGyE(Gray equivalent)/12Fx,55.2GyE/12Fx,56.4GyE/12Fx,57.6GyE/12Fx and 58.8GyE/12Fx ].
  Interventions: Radiation: carbon ion radiotherapy

INTERVENTIONS:
Radiation: carbon ion radiotherapy — dose escalation radiotherapy with five levels of dose from 54GyE/12Fx to 58.8GyE/12Fx

SUMMARY:
The arm of this study is to explore the optimal dose of 12 fractions of carbon ion radiotherapy for prostate cancer in our center.

DETAILED DESCRIPTION:
The radiation dose of 51.6GyE in 12 fractions is currently widely used in Japan, and clinical studies of 51.6GyE/12Fx have also been carried out for SBRT. There are some differences in equipment and carbon ion treatment planning system used between Japan and our center. Therefore, we designed this phase I clinical study to explore the optimal dose of 12 fractions of carbon ion radiotherapy for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of prostate
* Stage cT1-3N0M0 localized prostate cancer
* No lymph nodes or distant metastasis
* Age ≥ 45 and < 85 years of age
* Karnofsky Performance Score ≥70
* No previous pelvic radiation therapy (RT)
* No previous prostatectomy
* No previous invasive cancer (within 5 years before the prostate cancer diagnosis)
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* No pathologically confirmed adenocarcinoma of the prostate
* Pelvic lymph node metastasis (N1)
* Distant metastasis (M1)
* Previous pelvic radiotherapy
* Previous prostatectomy

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with prostate cancer
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months after the completion of CIRT
  Treatment related acute toxicity assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Biochemical failure free survival,bFFS | From the complation of CIRT,a median of 5 years
  The PSA less than nadir plus 2ng/ml
Overall survival | From the diagnosis of prostate cancer,a median of 5 years
  The time from diagnosis to death from any cause
Progression free survival | From the complation of CIRT,a median of 5 years
  The time from complation of CIRT to tumor progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No